CLINICAL TRIAL: NCT01305278
Title: The Efficacy of Balance Gaming as an Adjunct to Vestibular Rehabilitation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We unfortunately experienced recruitment difficulties with this study for the past few years.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, David Pothier, Assistant Professor, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHN-TGH-NO-0004
Record Dates: First submitted 2011-02-16; First posted 2011-02-28 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Vestibular Diseases; Disturbance; Balance, Labyrinth
Keywords: Balance; Rehabilitation; Vestibular
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): No Wii balance gaming undertaken
- Wii during vestibular rehab only (Active Comparator): To start Wii Balance Gaming from the beginning of vestibular rehabilitation.
  Interventions: Other: Use of Nintendo Wii Balance Gaming system
- Wii whilst on waiting list and rehab (Active Comparator): Wii Balance Gaming whilst on waiting list for vestibular rehabilitation. To continue with Wii Balance Gaming until end of vestibular rehabilitation.
  Interventions: Other: Use of Nintendo Wii Balance Gaming system

INTERVENTIONS:
Other: Use of Nintendo Wii Balance Gaming system — Use of Nintendo Wii Balance Gaming system
  Other Names: Nintendo, Wii, Balance Board, Wii Fit
  Arms: Wii during vestibular rehab only; Wii whilst on waiting list and rehab

SUMMARY:
Patients with a unilateral vestibular loss often complain of dizziness and imbalance. Movement usually increases these symptoms often resulting in patients avoiding these movements, causing further limitations in their activities of daily living. Vestibular Rehabilitation (VR) involves a series of adaptation and balance exercises to improve symptoms of postural stability. There is evidence that stroke patients gain benefit in their rehabilitation from using gaming consoles (Nintendo Wii Balance) and we believe that similar advantages can be shown for balance patients. We plan a 3 arm study. As there is a considerable wait list for VR, the first arm will receive a Wii console and instructions to use it on the wait list and during VR. The second arm will receive a Wii console and instructions at the end of the waiting list and will use it during VR only and the control group will receive no Wii. All will spend the same time on the wait list and will receive identical assessments and VR

DETAILED DESCRIPTION:
None required

ELIGIBILITY:
Inclusion Criteria:

* Unilateral vestibular loss
* Uncompensated
* Present for >6 months

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Index | t=0 (at initial assessment)
  Dynamic Gait index assessed by questionnaire at initial assessment (t=0) and then at 6 (midway through wait list), 12 (beginning of vestibular rehabilitation) and 18 weeks (end of vestibular rehabilitation)
  All groups compared at baseline
Dizziness Handicap Index | t=6 weeks
  Dynamic Gait index assessed by questionnaire at initial assessment (t=0) and then at 6 (midway through wait list), 12 (beginning of vestibular rehabilitation) and 18 weeks (end of vestibular rehabilitation)
  Group 1 (Wii during wait list and Vestibular Rehab) compared to Group 3 (Control)
Dizziness Handicap Index | t=12 weeks
  Dynamic Gait index assessed by questionnaire at initial assessment (t=0) and then at 6 (midway through wait list), 12 (beginning of vestibular rehabilitation) and 18 weeks (end of vestibular rehabilitation)
  Group 1 (Wii during wait list and Vestibular Rehab) compared to Group 3 (Control)
  All groups compared as a baseline before Vestibular Rehab
Dizziness Handicap Index | t=18 weeks
  Dynamic Gait index assessed by questionnaire at initial assessment (t=0) and then at 6 (midway through wait list), 12 (beginning of vestibular rehabilitation) and 18 weeks (end of vestibular rehabilitation)
  Group 2 (Wii during Vestibular Rehab only) compared to Group 3 (Control)

SECONDARY OUTCOMES:
Modified Clinical Test of Sensory Interaction on Balance | t=0 (at initial assessment), t=6 weeks, t=12 weeks, t=18 weeks
  mCTSIB assessed by blinded assessor at initial assessment (t=0)and then at 12 (beginning of vestibular rehabilitation) and 18 weeks (end of vestibular rehabilitation)
Activity Specific Balance Confidence Scale | t=0 (at initial assessment), t=6 weeks, t=12 weeks, t=18 weeks
  Activity Specific Balance Confidence Scale assessed by questionnaire at initial assessment (t=0)and then at 6 (midway through wait list), 12 (beginning of vestibular rehabilitation) and 18 weeks (end of vestibular rehabilitation)
Dynamic Gait Index score | t=0 (at initial assessment), t=12 weeks, t=18 weeks
  Dynamic Gait index assessed by blinded assessor at initial assessment (t=0)and then at 12 weeks (beginning of vestibular rehabilitation) and 18 weeks (end of vestibular rehabilitation)

CONTACTS AND LOCATIONS:
Overall Officials: John A Rutka, MD FRCS(C), Principal Investigator — Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada